CLINICAL TRIAL: NCT01477398
Title: Improved Patient Recovery of Spontaneous Respiration After Anesthesia With Hypercapnic Hyperpnoea
Brief Title: Improved Patient Recovery After Anesthesia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 36354
Record Dates: First submitted 2011-11-14; First posted 2011-11-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Recovery From Anesthesia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inspired CO2 (Active Comparator): Inspired CO2
  Interventions: Device: QED-100
- No intervention: Standard of Care (No Intervention): tidal volume and respiratory rate are not changed during recovery from anesthesia

INTERVENTIONS:
Device: QED-100 — Use of the QED-100 results in mild hypercapnia during emergence
  Other Names: Quick Recovery Device; AneClear
  Arms: inspired CO2

SUMMARY:
The proposed study will measure the incidence of adverse events and the decrease in time to meet discharge criteria from the post anesthesia care unit when hypercapnic and hyperpnoea are used during emergence.

DETAILED DESCRIPTION:
Hypercapnia has been used in conjunction with hyperpnoea to provide a more rapid return of responsiveness after inhaled anesthesia. The benefits of accelerating patient recovery in the operating room may extend to the post anesthesia care unit if the patient is more alert and easier to care for when they arrive in the unit. Respiratory patterns and gas levels - including CO2, O2, and anesthetic vapor - will be measured in order to better understand a patient's respiratory status during recovery.

In Feb 2009 we finished our first study (IRB 26111) and submitted a publication. The journal reviewers identified a serious limitation: we could not report whether the treated patients recovered from anesthesia faster because the treatment (inspired CO2) caused them to breath more vigorously or because the treatment caused the anesthetic vapors to be cleared more rapidly from the brain. Our new application uses essentially the same study protocol as the former study but adds chest bands to measure the patient's rate of breathing and expired gas monitoring to measure the rate at which the vapors are removed.

ELIGIBILITY:
Inclusion Criteria:

* adult ASA class I-III subjects of both genders scheduled to undergo eye surgery at the Moran Hospital.

Exclusion Criteria:

* a history of renal or hepatic disease, chronic alcohol or drug abuse, disabling neuropsychiatric disorder, hypersensitivity, or unusual response to other halogenated anesthetics, pulmonary hypertension, increased intracranial pressure, seizure disorder, or personal/familial history of malignant hyperthermia, and current smokers.
* Subjects will also be excluded if they are currently being treated with known hepatic enzyme-inducing drugs (e.g., phenobarbital, dilantin, or isoniazid) or with drugs known to alter anesthetic requirements (e.g., opiates, clonidine, alpha2 agonists, alcohol, anticonvulsants, antidepressants, barbiturates, benzodiazepines or other tranquilizers).
* Subjects will also be excluded if they have intolerance to non-steroidal anti-inflammatories.
* In addition subjects who have received general anesthesia within the previous 7 days, received any investigational drug within the previous 28 days, or participated in a previous isoflurane or desflurane study will be excluded.
* Female subjects can be neither pregnant nor breast feeding.
* Subjects with significant restrictive lung disease will also be excluded.
* Subjects passing these criteria will be further evaluated with a medical history including medications, abbreviated physical examination, clinical laboratory tests (urine drug test), and a urine or serum human chorionic gonadotropin pregnancy test for women with childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
treatment (inspired CO2) caused patients to breath more vigorously | 30 min
  Chest bands measuring the patients tidal volume will show that patients who receive the treatment will have larger tidal volumes than patients in the control group during the first 10 minutes after the end of surgery

SECONDARY OUTCOMES:
treatment caused the anesthetic vapors to be cleared more rapidly | 30 min
  A anesthetic gas analyzer will measure the amount of anesthetic gas in the patient's exhaled gas and will show that patients who receive the treatment will have lower exhaled anesthetic gas concentration than patients in the control group during the first 10 minutes after the end of surgery